CLINICAL TRIAL: NCT06376253
Title: A Phase I, Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Dosimetry, and Preliminary Activity of [177Lu]Lu-EVS459 in Patients With Ovarian and Lung Cancers
Brief Title: A Phase I Study of [177Lu]Lu-EVS459 in Patients With Ovarian and Lung Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study termination based on sponsor decision due to lack of tolerability observed with [177Lu]Lu-EVS459
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGIZ943A12101; 2023-507674-41-00 (Other: CTIS)
Record Dates: First submitted 2024-04-02; First posted 2024-04-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Lung Cancer
Keywords: ovarian cancer; non-squamous non-small cell lung cancer (non sq. NSCLC); advanced solid tumors; radioligand therapy (RLT); [177Lu]Lu-EVS459; [68Ga]Ga-EVS459; folate receptor (FR)
MeSH Terms: conditions — Ovarian Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): Patients will receive [68Ga]Ga-EVS459 and, if eligible, [177Lu]Lu-EVS459
  Interventions: Drug: [68Ga]Ga-EVS459; Drug: [177Lu]Lu-EVS459

INTERVENTIONS:
Drug: [68Ga]Ga-EVS459 — Radioligand imaging agent
Drug: [177Lu]Lu-EVS459 — Radioligand therapy

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, dosimetry and preliminary efficacy of [177Lu]Lu-EVS459 and the safety and imaging properties of [68Ga]Ga-EVS459 in patients aged ≥ 18 years with advanced high-grade serous ovarian cancer (OC) or locally advanced unresectable or metastatic non-squamous non-small cell lung carcinoma (non-sq. NSCLC).

DETAILED DESCRIPTION:
The study will be done in two parts. The first part is called "escalation" and the second part is called "expansion". In both parts of the study, patients will initially be imaged with a [68Ga]Ga EVS459 positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI) scan. In the escalation part, different doses of [177Lu]Lu-EVS459 will then be tested to identify recommended dose(s) (RD(s)) for further evaluation. The expansion part of the study will examine the safety and preliminary efficacy of [177Lu]Lu-EVS459 at the RD(s) determined during the escalation part. The end of study will occur when at least 80% of the patients in the expansion part have completed the follow-up for disease progression or discontinued from the study for any reason, and all patients have completed treatment and the 36-month long-term follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Age >= 18 years old
* Patients with advanced high-grade serous ovarian cancer (OC) or locally advanced unresectable or metastatic non-squamous non-small cell lung cancer (non sq. NSCLC) with disease progression following, or intolerance to, at least 1 line of therapy

Key Exclusion Criteria:

* Absolute neutrophil count (ANC) < 1.5 x 10^9/L, hemoglobin < 10 g/dL, or platelet count < 100 x 10^9/L
* QT interval corrected by Fridericia's formula (QTcF) ≥ 470 msec
* Creatinine clearance < 60 mL/min
* Unmanageable urinary tract obstruction or urinary incontinence
* Radiation therapy within 4 weeks prior to the first dose of [177Lu]Lu-EVS459

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-09-08 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities of [177Lu]Lu-EVS459 | From start of study treatment until 6 weeks after
  A dose limiting toxicity (DLT) is defined as any adverse event or abnormal laboratory value of CTCAE (version 5.0) Grade 3 or higher that occurs within the DLT evaluation period and that is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications with a few exceptions defined in the study protocol. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Incidence and severity of adverse events and serious adverse events of [177Lu]Lu- EVS459 | From start of study treatment until completion of the 36 month follow up , assessed up to approximately 42 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) and through the monitoring of relevant clinical and laboratory safety parameters.
Dose modifications for [177Lu]Lu- EVS459 | From start of study treatment until last dose of study treatment, assessed up to approximately 24 weeks
  Dose modifications (dose interruptions and reductions) for [177Lu]Lu-EVS459 will be assessed and summarized using descriptive statistics. The number of patients with dose modification will be summarized by treatment groups.
Dose intensity for [177Lu]Lu- EVS459 | From start of study treatment until last dose of study treatment, assessed up to approximately 24 weeks
  Dose intensity for [177Lu]Lu- EVS459 will be assessed and summarized using descriptive statistics. Dose intensity is computed as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 42 months
  ORR is defined as the proportion of patients with a BOR of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.
Duration of Response (DOR) | Up to approximately 42 months
  DOR is the time between the first documented response (CR or PR) and the date of progression according to RECIST v1.1 guidelines.
Disease control rate (DCR) | Up to approximately 42 months
  DCR is defined as the proportion of patients with a BOR of CR, PR, or stable disease according to RECIST v1.1 guidelines.
Progression free survival (PFS) | Up to approximately 42 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression according to RECIST v1.1 guidelines or death due to any cause.
Area Under the Curve (AUC) of [177Lu]Lu-EVS459 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes and 30 minutes, 1, 2, 4, 6 and 12 hours), Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  The [177Lu]Lu-EVS459 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. AUC will be determined by non-compartmental methods.
Total body clearance of [177Lu[Lu-EVS459 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes and 30 minutes, 1, 2, 4, 6 and 12 hours), Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  The [177Lu]Lu-EVS459 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Total body clearance will be determined by non-compartmental methods.
Observed maximum plasma concentration (Cmax) of [177Lu]Lu-EVS459 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes and 30 minutes, 1, 2, 4, 6 and 12 hours), Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  The [177Lu]Lu-EVS459 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Cmax will be determined by non-compartmental methods.
Volume of distribution during the terminal phase following intravenous elimination (Vz) of [177Lu]Lu-EVS459 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes and 30 minutes, 1, 2, 4, 6 and 12 hours), Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  The [177Lu]Lu-EVS459 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Vz will be determined by non-compartmental methods.
Terminal elimination half-life (T1/2) of [177Lu]Lu-EVS459 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes and 30 minutes, 1, 2, 4, 6 and 12 hours), Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  The [177Lu]Lu-EVS459 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. T1/2 will be determined by non-compartmental methods.
Urinary excretion of radioactivity expressed as a percentage of injected activity (%IA) | Cycle 1: Pre-infusion, beginning of infusion to first SPECT/CT image acquisition, first SPECT/CT image acquisition and 6 hours post-end-of infusion(EOI), 6-24 hours post-EOI, 24-48 hours post-EOI, 48-72 hours post-EOI. The duration of a cycle is 6 weeks.
  Urine elimination data for [177Lu]Lu-EVS459 will be assessed based on decay-corrected urine radioactivity concentration data. Urine elimination data will be expressed as percentage of injected activity (%IA).
Renal clearance of [177Lu]Lu- EVS459 | Cycle 1: Pre-infusion, beginning of infusion to first SPECT/CT image acquisition, first SPECT/CT image acquisition and 6 hours post-end-of infusion(EOI), 6-24 hours post-EOI, 24-48 hours post-EOI, 48-72 hours post-EOI. The duration of a cycle is 6 weeks.
  Urine samples will be collected over specified time intervals and analysed for radioactivity. Renal clearance of 177Lu-EVS459 will be summarized using descriptive statistics.
Absorbed dose of [177Lu]Lu- EVS459 | Cycle 1 Day 1, Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  The absorbed dose in normal tissues and tumor lesions will be summarized with descriptive statistics.
  Lesion number will be assigned by dosimetry expert.
Time-activity curves (TACs) related to [177Lu]Lu-EVS459 uptake in organs and tumor lesions | Cycle 1 Day 1, Cycle 1 Day 2 (24 hours), Cycle 1 Day 3 (48 hours), Cycle 1 Day 4 (72 hours), Cycle 1 Day 8 (168 hours). The duration of a cycle is 6 weeks.
  Time-activity curves (TACs) for the various organs and tumor lesions will be produced as fraction of injected activity per gram of tissue (%IA/g) as a function of time.
Incidence and severity of adverse events and serious adverse events of [68Ga]Ga-EVS459 | From Imaging visit until 14 days after 68Ga-EVS459 administration or until first dose of study treatment, assessed up to approximately 14 days
  The distribution of adverse events will be done via the analysis of frequencies for treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) and through the monitoring of relevant clinical and laboratory safety parameters.
Visual and quantitative assessment of [68Ga]Ga-EVS459 uptake in normal tissues and tumor lesions over time | From 0 up to approximately 3 hours after [68Ga]Ga-EVS459 dosing
  After [68Ga]Ga-EVS459 administration, [68Ga]Ga-EVS459 PET/CT or PET/MRI will be performed. Standardized uptake values (SUVs) of [68Ga]Ga-EVS459 in normal tissues and tumor lesions over time will be summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.